CLINICAL TRIAL: NCT04045093
Title: Rationale and Design of Dabigatran for Mitral Stenosis Atrial Fibrillation Trial
Brief Title: Dabigatran for Mitral Stenosis Atrial Fibrillation
Acronym: David-MS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Chun Ka, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAMS-01
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation; Mitral Stenosis
MeSH Terms: conditions — Atrial Fibrillation; Mitral Valve Stenosis | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Intervention Model Description: Prospective study with randomization in 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dabigatran etexilate (Experimental): Subjects randomized into this group will be prescribed with either Dabigatran 150mg or Dabigatran 110mg (twice daily) according to creatinine clearance level) for stroke prevention.
  Interventions: Drug: Dabigatran etexilate
- Warfarin (Active Comparator): Subjects randomized into this group will be prescribed with Warfarin with dosage adjustment according to INR level (targeting to INR 2-3) for stroke prevention.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran etexilate — Subjects will be randomized into 2 groups in a 1:1 ratio, to receive either Dabigatran or Warfarin for stroke prevention, in a open-label design.
  Other Names: Pradaxa
  Arms: Dabigatran etexilate
Drug: Warfarin — Subjects will be randomized into 2 groups in a 1:1 ratio, to receive either Dabigatran or Warfarin for stroke prevention, in a open-label design.
  Arms: Warfarin

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrythmia encountered in clinical practice and patients suffer from this are at increased risk of ischemic stroke and systemic thromboembolism due to the formation and embolism of left atrial thrombi. Current international guidelines recommend non-vitamin K oral anticoagulants (NOACs) for stroke prevention amongst these patients with non-valvular atrial fibrillation (AF) at significant ischemic stroke risk, given the superior safety and comparable efficacy of NOACs over warfarin. However, the safety and efficacy of NOACs had not been evaluated in AF patients with underlying mitral stenosis (MS) thereby the currently recommended stroke prevention strategy remains warfarin therapy for AF patients with underlying MS. A local study is initiated to compare efficacy and safety of Dabigatran with Warfarin therapy in AF patients with moderate to severe MS.

DETAILED DESCRIPTION:
While the stroke risk amongst AF patients appears heterogeneous, patients with underlying valvular heart diseases, particularly MS, are at very high risk for stroke if left un-anticoagulated. However, this group of patients was typically excluded in randomized control trials. As a result, current international guidelines for management of AF do not recommend NOACs for stroke prevention in AF patients with underlying moderate or severe MS. Nonetheless off-label use of NOACs in patients with MS is not uncommon in the real world practice.

This is of particular importance for Asian AF patients, in whom MS remains relatively prevalent despite a declining trend. More importantly, the much higher baseline risk of intracranial haemorrhage and apparently higher ischemic stroke risk in Asian populations potentially undermine the benefits of Warfarin therapy. On the other hand, the efficacy and safety of NOACs compared with Warfarin appear to be even higher in Asian population than the non-Asian population as shown in sub-analyses pivotal randomised control trials as well as in the real world evidence. This study refers as a prospective, randomized, open-label trial with blinded end-point adjudication, aiming at evaluating the safety and efficacy of Dabigatran for stroke prevention in AF patients with underlying moderate or severe MS.

After providing written informed consent, study participants from participating local centres will be randomized into 2 groups in a 1:1 ratio, to receive either Dabigatran (150mg or 110mg according to creatinine clearance level, twice daily) or Warfarin (targeting in the international normalized ratio (INR) range 2-3) in an open-label design. In a year of individual study period, vital signs, laboratory blood check and adverse events will be monitored, and primary and secondary outcomes will be assessed. The estimated sample size is approximately 370 participants. On addition, a subgroup of patients up to 10% of the target sample size will be invited for an one-time non-invasive magnetic resonance imaging (MRI) for assessment of any intra-cardiac thrombus.

The results will be an important contribution to the stroke prevention strategy for patients with MS and may be immediately translatable to real clinical practice. Ultimately, this study will provide the necessary evidence for establishing universal guidelines for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation documented with standard 12-lead ECG documented atrial fibrillation on the day of screening or randomization
* Patients with age ≥ 18 years
* Patients with moderate or severe mitral stenosis, i.e. mitral valvular area (MVA) ≤ 2.5cm2
* Patients should be able to provide a written informed consent
* Patients should have all 4 inclusion-criteria fulfilled to be qualified for the study

Exclusion Criteria:

* Patients with mechanical prosthetic valve, or with active endocarditis
* Patients with planned valvular intervention within 1 year
* Patients with left atrial appendage occlusive device
* Patients with planned AF ablation
* Unexplained anemia (haemoglobin level < 10g/dL) or thrombocytopenia (platelet count < 100x10*9/L)
* Need for anticoagulant therapy of disorders other than atrial fibrillation
* Patients receiving antiplatelet therapy for disorders other than atrial fibrillation
* Uncontrolled hypertension (systolic blood pressure > 180mmHg and/or diastolic blood pressure > 100mmHg)
* Estimated creatinine clearance ≤ 30mL/min
* Liver dysfunction of Child Pugh stage B or C
* Women who are pregnant or of childbearing potential who refuse to use a medically acceptable form of contraception throughout the study
* Patients considered unreliable by the investigator or have a life expectancy less than 1 year because of concomitant disease, or has any condition, which in the opinion of the investigator, would not allow safe participation in the study (e.g. drug addiction, alcohol abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite of stroke, systemic embolism, myocardial infarction, and death from cardiovascular or unknown cause. | 1 year
  Stroke is classified into ischemic or hemorrhagic stroke, as confirmed by computed tomography or magnetic resonance imaging.
  Systemic embolism is defined as an acute vascular occlusion of an extremity or organ other than the brain, documented by imaging, surgery, and/or autopsy.
  Myocardial infarction is defined according to the latest ACC/AHA/ACEP/NAEMSP/SCAI guideline for the management of patients with acute coronary syndromes, with the assessment of electrocardiography, cardiac troponin values and presence of symptoms.
  Death is counted when subject is medically certified of death, resulted from cardiovascular or unknown cause.

SECONDARY OUTCOMES:
Ischemic stroke | 1 year
  It is defined as the first episode during follow-up of new-onset of neurological symptoms attributable to a cerebral infarct, as confirmed by computed tomography or magnetic resonance imaging, lasting more than 24 hours.
Hemorrhagic stroke | 1 year
  It is defined as the first episode during follow-up of new-onset of neurological symptoms attributable to an intraparenchymal or subarachnoid hemorrhage, as confirmed by computed tomography or magnetic resonance imaging.
Systemic embolism | 1 year
  It is defined as an acute vascular occlusion of an extremity or organ other than the brain, documented by imaging, surgery, and/or autopsy.
Major bleeding | 1 year
  Bleeding being categorized as BARC type 3 or higher is regarded as major bleeding.
Death | 1 year
  It is counted when subject is medically certified of death.

CONTACTS AND LOCATIONS:
Overall Officials: Siu Han Jo Jo Hai, Bachelor, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong / Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request to the corresponding author

REFERENCES:
- [Derived] Zhou M, Chan EW, Hai JJ, Wong CK, Lau YM, Huang D, Lam CC, Tam CCF, Wong YTA, Yung SYA, Chan KWK, Feng Y, Tan N, Chen JY, Yung CY, Lee KL, Choi CW, Lam H, Ng A, Fan K, Jim MH, Yiu KH, Yan BP, Siu CW. Protocol, rationale and design of DAbigatran for Stroke PreVention In Atrial Fibrillation in MoDerate or Severe Mitral Stenosis (DAVID-MS): a randomised, open-label study. BMJ Open. 2020 Sep 25;10(9):e038194. doi: 10.1136/bmjopen-2020-038194. PMID 32978200